CLINICAL TRIAL: NCT00085410
Title: Phase II and Pharmacodynamic Study of PS-341 in Patients With Unresectable or Metastatic Adenocarcinoma of the Bile Duct or Gallbladder
Brief Title: Bortezomib in Treating Patients With Unresectable Locally Advanced or Metastatic Adenocarcinoma of the Bile Duct or Gallbladder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was discontinued early due to no confirmed partial responses.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00046; NCI-2009-00046 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000369715; 03-042; 03-042 (Other: Fox Chase Cancer Center); 6135 (Other: CTEP)
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Adenocarcinoma of the Extrahepatic Bile Duct; Adenocarcinoma of the Gallbladder; Advanced Adult Primary Liver Cancer; Gastrointestinal Cancer; Localized Unresectable Adult Primary Liver Cancer; Recurrent Adult Primary Liver Cancer; Recurrent Extrahepatic Bile Duct Cancer; Recurrent Gallbladder Cancer; Unresectable Extrahepatic Bile Duct Cancer; Unresectable Gallbladder Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms; Carcinoma, Hepatocellular; Bile Duct Neoplasms; Gallbladder Neoplasms | interventions — Bortezomib

ARMS (1):
- Arm I (Experimental): Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11.
  Interventions: Drug: bortezomib

INTERVENTIONS:
Drug: bortezomib — Given IV

SUMMARY:
This phase II trial is studying how well bortezomib works as first-line systemic therapy in treating patients with unresectable locally advanced or metastatic adenocarcinoma (cancer) of the bile duct or gallbladder. Bortezomib may stop the growth of tumor cells by blocking the enzymes necessary for their growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the objective response rate in patients with unresectable locally advanced or metastatic adenocarcinoma of the bile duct or gallbladder treated with bortezomib.

SECONDARY OBJECTIVES:

I. Determine the time to disease progression in patients treated with this drug.

II. Determine the overall survival of patients treated with this drug. III. Correlate the degree of proteasome inhibition in peripheral blood with degree of proteasome inhibition in tumor specimens of patients treated with this drug.

IV. Correlate phenotypic expression of NF-kB, p53, and other molecular markers in biliary washings and tumor biopsies with clinical outcomes in patients treated with this drug.

V. Correlate treatment with this drug with changes in phenotypic expression of molecular markers in these patients.

OUTLINE: This is an open-label, multicenter study.

Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Absolute neutrophil count >= 1,500/mm3
* No psychiatric illness or social situation that would preclude study compliance
* Chemotherapy administered solely as a radiosensitizer or as adjuvant therapy and investigational or targeted therapies (i.e., inhibitors of the epidermal growth factor receptor) will not count toward the maximum of 2 prior regimens allowed
* Histologically or cytologically confirmed adenocarcinoma of the intrahepatic or extrahepatic bile duct or gallbladder:

  * Locally advanced or metastatic disease
* At least 1 unidimensionally measurable lesion >=20 mm by conventional techniques OR >= 10 mm by spiral CT scan
* Not amenable to curative surgical resection
* No known brain metastases
* Performance status:

  * ECOG 0-2
* Life expectancy:

  * More than 12 weeks
* Platelet count >= 100,000/mm3
* WBC >= 3,000/mm3
* AST and ALT ≤ 2.5 times upper limit of normal (ULN) [Note: Biliary shunting or stenting allowed to achieve the required bilirubin and transaminase levels]
* Bilirubin ≤ 1.5 times ULN [Note: Biliary shunting or stenting allowed to achieve the required bilirubin and transaminase levels]
* Creatinine within ULN OR Creatinine clearance >= 60 mL/min
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No symptomatic cardiac arrhythmia within the past 4 weeks
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No underlying neuropathy >= grade 2
* No history of allergic reaction to boron, mannitol, or bortezomib
* No active or ongoing infection
* No concurrent uncontrolled illness
* No medical or psychiatric condition that would preclude study participation
* No prophylactic granulocyte or platelet growth factors (filgrastim [G-CSF] or sargramostim [GM-CSF])
* Prior chemotherapy as a radiosensitizer (e.g., fluorouracil or gemcitabine) with radiotherapy is allowed as adjuvant therapy after resection for locally advanced disease provided there is evidence of disease progression
* No more than 2 prior chemotherapy regimens for locally advanced or metastatic disease
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent anticancer agents or therapies
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-01; Primary Completion 2008-08 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Cohen, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Denlinger CS, Meropol NJ, Li T, Lewis NL, Engstrom PF, Weiner LM, Cheng JD, Alpaugh RK, Cooper H, Wright JJ, Cohen SJ. A phase II trial of the proteasome inhibitor bortezomib in patients with advanced biliary tract cancers. Clin Colorectal Cancer. 2014 Jun;13(2):81-6. doi: 10.1016/j.clcc.2013.12.005. Epub 2014 Jan 4. PMID 24512954

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through physician referral at: Fox Chase Cancer Center. The trial was discontinued early due to no confirmed partial responses.
Pre-assignment Details: Twenty individuals were enrolled in this study over a four year period.
Period: Overall Study
Arm/Group | Arm I
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm I
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 20
Site of Primary Tumor [Number; unit: participants]
  Gallbladder | 6
  Intrahepatic or extrahepatic cholangiocarcinoma | 14
Site of Metastases [Number; unit: participants] — Multiple Metastases possible per patient
  participants
    Liver | 14
    Lymph nodes | 7
    Lung | 5
    Other | 2
Eastern Cooperative Oncology Group Performance Status [Number; unit: participants] — Grade 0: Fully active, able to carry on all pre-disease performance without restriction
  Grade 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature
  participants
    Grade 0 | 7
    Grade 1 | 13
Previous Treatment [Number; unit: participants]
  None | 10
  Chemotherapy only | 4
  Chemotherapy/radiation therapy | 5
  Other | 1
Previous Surgery [Number; unit: participants]
  Yes: Cholecystectomy | 4
  Yes: Liver section | 1
  No | 15

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Objective Response Rate (ORR) was determined by best response on radiologic assessment (computed tomography or magnetic resonance imaging) according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.0.
Time Frame: Up to 1 year
Population: Per protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 20
Participants
  Stable Disease | 10
  Partial Response (Unconfirmed) | 1
  Progressive Disease | 8
  Withdrew Consent Before Evaluation | 1

2. Secondary Outcome: Time to Disease Progression
Description: Time from initiation of therapy to first progressive disease.
Time Frame: Up to 1 year
Population: 1 patient who withdrew consent prior to the first disease evaluation was excluded.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I
Number analyzed (Participants) | 19
months | 5.8 [0.7 to 77.6]

3. Secondary Outcome: Overall Survival
Description: The time from initiation of therapy to death or last follow-up.
Time Frame: Up to 1 year
Population: 1 patient who withdrew consent prior to the first disease evaluation was excluded.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I
Number analyzed (Participants) | 19
months | 9 [4.6 to 18.5]

4. Secondary Outcome: Correlation of the Degree of Proteasome Inhibition in Peripheral Blood With the Degree of Proteasome Inhibition in Tumor Specimens
Description: Proteasome inhibition compared between tumor specimens and peripheral blood. Sufficient tissue samples are required for this analysis.
Time Frame: Once in the screening period (within 14 days of starting treatment)
Population: Insufficient amount of patient samples collected for analysis
Arm/Group | Arm I
Number analyzed (Participants) | 0

5. Secondary Outcome: Correlation of Phenotypic Expression of NF-kB, p53, and Other Molecular Markers in Biliary Washings and Tumor Biopsies With Clinical Outcomes
Description: Evaluation of clinical outcomes with expression of molecular markers specified and others. Sufficient amount of biliary washings and tumor biopsies needed for analysis.
Time Frame: Once in the screening period (within 14 days of starting treatment)
Population: Insufficient amount of patient samples collected for analysis
Arm/Group | Arm I
Number analyzed (Participants) | 0

6. Secondary Outcome: Correlation of Treatment With Changes in Phenotypic Expression of Molecular Markers
Description: Phenotypic expression of molecular markers before and after study treatment
Time Frame: Duration of study treatment
Population: Insufficient amount of patient samples collected for analysis
Arm/Group | Arm I
Number analyzed (Participants) | 0

7. Post Hoc Outcome: Clinical Benefit Rate
Description: Best response to study treatment was confirmed complete response, partial response, or stable disease. Unconfirmed partial response was not included. The outcome measure data table is stratified into patients who a) received prior therapy b) did not receive prior therapy.
Time Frame: Up to 1 year
Population: 1 patient who withdrew consent prior to the first disease evaluation was excluded.
Measure: Number; unit: percentage of patients
Arm/Group | Arm I
Number analyzed (Participants) | 19
percentage of patients
  Patients who received prior therapy | 21
  Patients who did not receive prior therapy | 32

8. Post Hoc Outcome: 6-Month Survival
Description: The time from initiation of therapy to 6 months beyond.
Time Frame: 6 months
Population: 1 patient who withdrew consent prior to the first disease evaluation was excluded.
Measure: Number; unit: percentage of patients
Arm/Group | Arm I
Number analyzed (Participants) | 19
percentage of patients | 70

9. Post Hoc Outcome: 1-year Survival
Description: The time from initiation of initiation of therapy to 1 year beyond.
Time Frame: 1 year
Population: 1 patient who withdrew consent prior to the first disease evaluation was excluded.
Measure: Number; unit: percentage of patients
Arm/Group | Arm I
Number analyzed (Participants) | 19
percentage of patients | 38

10. Post Hoc Outcome: 6-Month and 1-Year Survival for Patients Who Derived Clinical Benefit From Study Treatment
Description: The time from initiation of therapy to 6 months beyond. Only patients who derived benefit from study treatment (stable disease, partial response, or complete response was best response) were included.
Time Frame: Up to 1 year
Population: Patients who derived benefit from study treatment (stable disease, partial response, or complete response was best response)
Measure: Number; unit: percentage of patients
Arm/Group | Arm I
Number analyzed (Participants) | 10
percentage of patients
  6-Month Survival | 90
  1-Year Survival | 69

11. Post Hoc Outcome: 6-Month and 1-Year Survival: Patients Who Did Not Derive Clinical Benefit From Study Treatment
Description: The time from initiation of therapy to 6 months beyond. Only patients who did not derive clinical benefit from study treatment (progressive disease or unconfirmed partial response was best response) were included.
Time Frame: Up to 1 year
Population: Patients who did not derive clinical benefit from study treatment (progressive disease was best response) only.
Measure: Number; unit: percentage of patients
Arm/Group | Arm I
Number analyzed (Participants) | 9
percentage of patients
  6-Month Survival | 44
  1-Year Survival | 11

ADVERSE EVENTS:
Arm/Group | Arm I
Serious Adverse Events (participants affected / at risk) | 4/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=20)
aseptic vasculitis (Nervous system disorders) | 1 (1)
cerebrovascular accident (Vascular disorders) | 1 (1)
meningitis (Nervous system disorders) | 1 (1)
renal insufficiency (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=20)
Anemia (Blood and lymphatic system disorders) | 15
Leukopenia (Blood and lymphatic system disorders) | 5
Neutropenia (Infections and infestations) | 5
thrombocytopenia (Skin and subcutaneous tissue disorders) | 14
Dehydration (Gastrointestinal disorders) | 3
dizziness (Nervous system disorders) | 4
Edema (General disorders) | 5
Elevated alkaline phosphatase (Metabolism and nutrition disorders) | 3
Elevated AST/ALT (Metabolism and nutrition disorders) | 7
Elevated creatinine (Metabolism and nutrition disorders) | 3
Fatigue (General disorders) | 18
GI obstruction (Gastrointestinal disorders) | 0
Hyperbilirubinemia (Metabolism and nutrition disorders) | 4
Hypertension (Cardiac disorders) | 4
Nausea (Gastrointestinal disorders) | 11
Pain (all sites) (General disorders) | 9
Rash/ulceration (Skin and subcutaneous tissue disorders) | 4
Sensory neuropathy (Nervous system disorders) | 6
Vomiting (Gastrointestinal disorders) | 7

LIMITATIONS AND CAVEATS:
The trial was discontinued early due to no confirmed partial responses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less